CLINICAL TRIAL: NCT07316387
Title: Neurobehavioral Development in Toddlers and Preschoolers in Relation to Prenatal Exposure of Mild Analgesics
Brief Title: Neurobehavioral Development in Toddlers and Preschoolers in Relation to Prenatal Exposure of Mild Analgesics (NeuroToP - a COPANA Follow up)
Acronym: NeuroToP
Status: Enrolling by invitation | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Casper Hagen, Associate Professor, Rigshospitalet, Denmark
Other Study IDs: COPANA_NEUROTOP
Record Dates: First submitted 2025-03-17; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Gonad Regulating Hormone Adverse Reaction; Analgesic Adverse Reaction; Developmental Disability; Adhd; Autism Spectrum Disorder; Language Development
MeSH Terms: conditions — Developmental Disabilities; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples Urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Healthy children originally recruited specifically for COPANA will be reinvited for follow up, including a child examination.
- The mothers and fathers of the children: The parents, i.e., the mother and father, of the healthy children. The parents will answer the inventories regarding the neurobehavioral development of the child and the general health questionnaire including parental educational level etc.

SUMMARY:
Fundamental aspects of both neurological and reproductive function are established in fetal life, and there is a present increased awareness of the potential effects of fetal exposures on neurodevelopmental and reproductive health of offspring. Experimental and epidemiological research studies strongly suggest that paracetamol and NSAID are endocrine disruptive in the fetus, which could increase the risks of some neurodevelopmental, reproductive, and urogenital disorders. In recent years, there has been an increasing rate of neurodevelopmental disorders such as ADHD and autism. The original cohort, the Copenhagen Analgesic Study (COPANA), is the first prospective human study designed primarily to assess the effect of fetal exposure to mild analgesics on male and female reproductive function. If the same children are examined with relevant neurobehavioral testing during mid-childhood, the study design allows the investigators to assess the effect of mild analgesics as well as other EDCs on neurodevelopmental health.

DETAILED DESCRIPTION:
Detailed Description In Denmark, mild analgesics such as acetaminophen (e.g. paracetamol) and non-steroidal anti-inflammatory drugs, NSAIDs (e.g. ibuprofen and acetylsalicylic acid), are sold over the counter, and up to 56% of pregnant women use mild analgesics during pregnancy. In vivo, in vitro, and ex vivo studies have shown that paracetamol directly perturbs hormone-dependent processes, which leads to disrupted reproductive development and neurodevelopment in both sexes. Fetal exposure in rodents has been shown experimentally to cause reproductive disorders of the male urogenital tract, including abnormalities in testicular function, sperm abnormalities, and sexual behavior. Experiments have shown disruption of female ovarian development resulting in reduced oocyte number and subsequent early ovarian insufficiency and reduced fertility. Fetal paracetamol exposure has been demonstrated to induce changes in neurotransmission in the brain manifesting in altered cognitive function, behavior, and locomotion. The studies have shown that the effect of paracetamol is dependent on the timing of exposure in relation to specific developmental processes, duration, and dose.

Population-based cohort studies have reported associations of prenatal exposure to EDCs and language development, autism spectrum disorder scores, as well as externalizing and internalizing behavior scores. Phthalates are one example of an endocrine disrupter used in a variety of consumer products. Human studies suggest an association between phthalate exposure and cognitive development. However, adverse effects of the recently introduced phthalate substitutes have only been sparsely studied, which will be a focus point in this study.

Animal studies suggest deleterious effects of fetal exposure to mild analgesics on both male and female gonadal development. In rodents, paracetamol administered in a single daily dose of 350 mg/kg at 13.5-21.5 days post coitum (dpc) was associated with reduced prostaglandin synthesis and delayed transition from germ cell mitosis to meiosis, causing fetal germ cell apoptosis in both female and male gonads. The long-term consequence seems to be most severe in the female, who becomes unable to form germ cells postnatally. In two studies, female offspring of mice treated with mild analgesics at 7 dpc to delivery and 13.5-21.5 dpc were born with reduced ovarian weight and with a 40-50% reduction in number of follicles. In adulthood, exposed animals gave birth to fewer pups per litter compared with controls.

Use of acetylsalicylic acid (150-250 mg/kg/day) in early and mid-pregnancy (dpc 13-21) has shown to be antiandrogenic, causing shorter AGD and decreased testosterone production in rodents. Furthermore, studies of rodents suggest that in both males and females, adverse reproductive effects are passed on to the next generations, indicating altered and inherited programming of the genome, i.e., epigenetic. Effects on fetal germ cell development with therapeutically relevant concentrations of analgesics have been confirmed in various experimental animal models.

Other medications, such as glucocorticoids and azoles, have previously been suggested to affect fetal germ cell development and will therefore also be incorporated in this study to adjust for possible effects when analyzing final data. Aniline is an organic compound found in many industrial products, pesticides, rubber, textiles, and tobacco smoke. The general population is inevitably exposed to aniline in daily life, and in vivo aniline is converted to paracetamol. In fact, studies have shown that paracetamol can be measured in urine samples of the general human population even with no prior intake of paracetamol, and similar to paracetamol, aniline has shown to exhibit similar anti-androgenic effects in male mice.

To date, no prospective human studies have assessed the effect of analgesic exposure on neurobehavioral development. COPANA is the first prospective human study designed primarily to assess the effect of fetal exposure to mild analgesics on male and female reproductive function. By inviting the same families to participate in the present study, unique information about essential prenatal exposure patterns of analgesics as well as other potential EDCs (e.g., fungicides and phthalates) is already available. Furthermore, essential parameters for the gonadal function of the children have been established in the previous study. These parameters can be directly included in analyses of associations to neurobehavioral development.

The primary objective of this study is to evaluate whether analgesic exposure during fetal life affects neurodevelopmental health in male and female toddlers and preschool children. Prenatal exposure to other potential endocrine-disrupting chemicals (e.g., fungicides and phthalates) on brain development will also be assessed. The families will be asked to complete inventories designed and validated to evaluate language development, ADHD and autism-like behavior, and gender-typical behavior-disorders that are more prevalent in gender-incongruent children and possibly linked with hormone-mediated brain development.

To elucidate underlying mechanisms, the study includes an analysis of the children's epigenetic profile and genetic variation in specific genes/promoter regions affecting prostaglandin action in parents, boys, and girls.

ELIGIBILITY:
Inclusion Criteria:

- Participant in the COPANA project

Exclusion Criteria:

* Premature birth
* Postterm birth
* Twin birth (gemelli)
* Severe disease in the child
* Stillbirth
* Late abortion

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is a population based prospective cohort study of 685 families (healthy pregnant mothers, biological fathers and their healthy male/female offspring.)There are two groups of participants in this study: 1. Healthy children recruited in 2020-2022 in the COPANA study and the parents, i.e. the mother and father, of the healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 685 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2028-05-27 (Estimated); Study Completion 2028-05-27 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P) (male and female children) | 2-5 years of age
  Parents will complete the BRIEF-P to assess their child's executive functioning, and the Global Executive Composite score will be used in the analysis.
BRIEF-P Global Executive Composite (GEC) (male and female children) | 2-5 years of age
  The Global Executive Composite (GEC) score is derived from the BRIEF-P questionnaire, which includes 63 items assessing executive functioning in preschool-aged children. The GEC score reflects the overall level of executive function difficulties and is calculated from the five clinical subscales: Inhibit, Shift, Emotional Control, Working Memory, and Plan/Organize.
BRIEF-P Emergent Metacognition Index (male and female children) | 2-5 years
  The EMI score reflects the child's ability to sustain ideas and activities in working memory and to plan and organize problem-solving approaches. It is composed of the Working Memory and Plan/Organize subscales and is critical for developing systematic metacognitive strategies.
Child Behavioral and Emotional Functioning - Child Behavior Checklist (CBCL) - (male and female children) | 2-5 years of age
  Behavioral and emotional functioning will be assessed using the Child Behavior Checklist (CBCL), a validated parent-report questionnaire. The CBCL provides a Total Score as well as multiple subscale scores reflecting specific behavioral and emotional domains. The questionnaire is completed electronically by the child's mother or father when the child is between 2 and 4 years of age.
  Unit of Measure: CBCL standardized score (T-score)
CBCL Total Problem Score (TPS) (male and female children) | 2-5 years of age
  The Total Problem Score (TPS) from the Child Behavior Checklist for Ages 1½-5 (CBCL/1½-5) is derived by summing responses of all items. The possible TPS ranges from 0 to 200, with higher scores representing more severe behavioral and emotional problems. According to standardized CBCL norms. Raw scores are converted to age- and sex-adjusted T-scores for interpretation.
CBCL Internalizing Score (male and female children) | 2-5 years of age
  The Internalizing Score is based on 24 items assessing emotional symptoms such as anxiety, depression, and withdrawal. The score range is 0-48.
CBCL Externalizing Score (male and female children) | 2-5 years of age
  The Externalizing Score is based on 36 items assessing behaviors such as aggression and rule-breaking. The score range is 0-72.
Danish MacArthur-Bates Communicative Development Inventories (MB-CDI) (male and female children) | 2-4 years
  Using the validated Danish MacArthur-Bates Communicative Development Inventories (MB-CDI) "Words and Sentences", which consists of a vocabulary check list (part I) and questions regarding sentences and grammar (part II). Distributed electronically to the mother of the child at age 2-4 years.
MB-CDI Vocabulary Size (Words Understood and Produced) (male and female children) | 2-4 years
  Assessed using Part I of the validated Danish version of the MacArthur-Bates Communicative Development Inventories (MB-CDI) "Words and Sentences". This section consists of a vocabulary checklist completed by the child's mother.
  Unit of Measure: Number of words understood and/or produced
MB-CDI Sentence and Grammar Use (male and female children) | 2-4 years of age
  Assessed using Part II of the Danish MB-CDI "Words and Sentences", which includes questions about the child's use of sentences and grammatical structures. The questionnaire is distributed electronically to the mother.
  Unit of Measure: Parental report of sentence complexity and grammatical usage (qualitative and/or categorical scoring)
Preschool Activities Inventory - Gender-typical behavior (male and female children) | 3-5 years
  Using the "Preschool Activities Inventory "(PSAI). This includes 24 items about the child's toy and activity preferences. The inventory holds 12 typical masculine and 12 typical feminine activities. The parents will score each activity on a likert scale which creates a composite score on the childs preferences.
Attention deficit hyperactivity disorder (ADHD) symptom load - Measured by the ADHD Rating Scale (male and female children) | At 5 years of age
  The ADHD Rating Scale (ADHD-RS) assesses ADHD symptom severity based on 26 items rated on a 4-point scale (0 = never, 3 = very often). The total score ranges from 0 to 78, with higher scores indicating greater symptom severity. The total score is calculated by summing all item scores.
Inattention symptom load - Measured by the ADHD Rating Scale (male and female children) | 5 years of age
  The ADHD Rating Scale Inattention Subscore is based on 9 items rated on a 4-point scale (0 = never, 3 = very often). Scores range from 0 to 27, with higher scores indicating greater severity of inattention symptoms.
Hyperactivity/Impulsivity symptom load - Measured by the ADHD Rating Scale (male and female children) | 5 years of age
  The ADHD Rating Scale Inattention Subscore is based on 9 items rated on a 4-point scale (0 = never, 3 = very often). Scores range from 0 to 27, with higher scores indicating greater severity of inattention symptoms.
Total Difficulties Score derived from the "Strengths and Difficulties Questionnaire" (SDQ) (male and female children) | 2-5 years
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item behavioral screening tool that assesses emotional and behavioral problems in children. The Total Difficulties Score is calculated by summing four subscales: Emotional Symptoms, Conduct Problems, Hyperactivity-Inattention, and Peer Problems (20 items in total). The Total Difficulties Score ranges from 0 to 40, with higher scores indicating greater emotional and behavioral difficulties. According to standardized norms, scores can be interpreted depending on age- and sex-specific cutoffs. The SDQ also includes a separate Prosocial Behavior subscale, which is not included in the Total Difficulties Score.

SECONDARY OUTCOMES:
Gross motor development (Parent reported) | 1-2 year
  Gross motor development will be assessed through parent-reported milestone data collected via a general health questionnaire.
  Units: months
Childhood Infections (Parent-Reported and Registry-Based Assessment) | 1-6 years old
  Infectious disease history during early childhood will be assessed using two sources:
  1. A general health questionnaire completed by the child's parent, covering frequency and type of infections.
  2. Clinical data extracted from the Danish electronic health record system Sundhedsplatformen, including diagnostic codes and treatment records related to infections.
  The combined data will be used to characterize infection burden, including number of infections, type (e.g., respiratory, gastrointestinal), and need for medical treatment.
Length (male and female children) | 2-4 years
  Length measured in centimeters.
Weight (male and female children) | 2-4 years
  Weight measured in kilograms
Head circumference (male and female children) | 2-4 years
  Head circumference measured in centimenters with measurement tape.
Waist circumference (male and female children) | 2-4 years
  Waist circumference measured in centimenters with measurement tape.
Hip circumference (male and female children) | 2-4 years
  Hip circumference measured in centimenters with measurement tape.
Digit length (male and female children) | 2-4 years
  2. and 4. finger length measured in milimeters with a caliper
Biceps skinfold (male and female children) | 2-4 years
  Skinfold measured above the biceps, measured in milimeters (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Triceps skinfold (male and female children) | 2-4 years
  Skinfold measured above the triceps, measured in milimeters (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Scapula skinfold (male and female children) | 2-4 years
  Skinfold measured above the flank, measured in milimeters Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Serum concentration of brain-derived neurotrophic factor (BDNF) (male and female children) | 2-4 years
  Serum concentration of brain-derived neurotrophic factor (BDNF) measured in ng/ml by using ELISA
Serum concentration of progesterone (male and female children) | 2-4 years
  Serum progesterone measured in nmol/L by using LC/MS-MS
Serum concentration of dehydroepiandrosterone (DHEA) (male and female children) | 2-4 years
  Serum concentration of dehydroepiandrosterone (DHEA) measured in nmol/L by using LC/MS-MS
Serum concentration of 17-hydroxypregnenolone (male and female children) | 2-4 years
  Serum concentration of 17-hydroxypregnenolone measured in nmol/L by using LC/MS-MS
Serum concentration of dihydroxytestosterone (male and female children) | 2-4 years
  Serum concentration of dihydroxytestosterone measured in nmol/L by using LC/MS-MS
Serum concentration of 11-deoxycorticosterone (male and female children) | 2-4 years
  Serum concentration of 11-deoxycorticosterone measured in nmol/L by using LC/MS-MS
Serum concentration of 17α-hydroxyprogesterone (male and female children) | 2-4 years
  Serum concentration of 17α-hydroxyprogesterone measured in nmol/L by using LC/MS-MS
Serum concentration of androstenedione (male and female children) | 2-4 years
  Serum concentration of the hormone androstenedione measured in nmol/L by using LC/MS-MS.
Serum concentration of 11-deoxycortisol (male and female children) | 2-4 years
  Serum concentration of 11-deoxycortisol measured in nmol/L by using LC/MS-MS
Serum concentration of corticosterone (male and female children) | 2-4 years
  Serum concentration of corticosterone measured in nmol/L by using LC/MS-MS
Serum concentration of 21-deoxycortisol (male and female children) | 2-4 years
  Serum concentration of 21-deoxycortisol measured in nmol/L by using LC/MS-MS
Serum concentration of cortisol (male and female children) | 2-4 years
  Serum concentration of cortisol measured in nmol/L by using LC/MS-MS
Serum concentration of cortisone (male and female children) | 2-4 years
  Serum concentration of cortisone measured in nmol/L by using LC/MS-MS
Serum concentration of aldosterone (male and female children) | 2-4 years
  Serum concentration of aldosterone measured in nmol/L by using LC/MS-MS
Serum concentration of dehydroepiandrosterone sulfate (DHEAS) (male and female children) | 2-4 years
  Serum concentration of dehydroepiandrosterone sulfate (DHEAS) measured in nmol/L by using LC/MS-MS
Serum concentration of IGF-binding protein 3 (male and female children) | 2-4 years
  Serum concentration of IGF-binding protein 3 measured in μg/L by using chemiluminescence Immunoassay
Serum concentration of anti-müllerian hormone (AMH) (male and female children) | 2-4 years
  Serum concentration of anti-müllerian hormone (AMH) measured in pmol/L using chemiluminescence Immunoassay
Serum concentration of estrone sulfate (male and female children) | 2-4 years
  Serum concentration of estrone sulfate measured in nmol/L by using LC/MS-MS
Serum concentration of luteinizing hormone (male and female children) | 2-4 years
  Serum concentration of luteinizing hormone (LH) measured in IU/L by chemiluminescence immunoassay
Serum concentration of Insulin-like growth factor-I (male and female children) | 2-4 years
  Serum concentration of Insulin-like growth factor-I measured in μg/L by using chemiluminescence Immunoassay
Serum concentration of Sex hormone Binding Globulin (SHBG) (male and female children) | 2-4 years
  Serum concentration of Sex hormone Binding Globulin (SHBG) measured in nmol/L by using hemiluminescence Immunoassay
Serum concentration of estradiol (male and female children) | 2-4 years
  Serum concentration of estradiol measured in pmol/L by using LC/MS-MS
Serum concentration of inhibin B (male and female children) | 2-4 years
  Serum concentration of inhibin B. The concentration will be measured by using the enzyme-linked immunosorbent assay. The unit nanogram/liters is found by dividing the weight of the product in nanograms with the volume of the product in liters.
Serum concentration of testosterone (male and female children) | 2-4 years
  Serum concentration of testosterone measured in nmol/L by using liquid chromatography tandem mass spectrometry (LC/MS-MS).
Serum concentration of follicular stimulating hormone (FSH) (male and female children) | 2-4 years
  Serum concentration of follicular stimulating hormone (FSH) measured in IU/L by chemiluminescence immunoassay
Flank skinfold (male and female children) | 2-4 years
  Skinfold measured above the flank, measured in milimeters (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Medical history (mother) | 2-4 years
  Medical history (mother) Retrieved from the digital journal system "Sundhedsplatformen"
Medical history (male and female children) | 2-4 years
  Retrieved from the digital journal system "Sundhedsplatformen" and from the health questionnaire distributed via Eboks.
Testes volumen (male children) | 2-4 years
  Ultrasound will be used to determine length, cross section and width of the testis measured in milimeters. Volume is calculated by multiplying length, cross section and width of the testes and we will report the volume in mm^3.
Testes volumen (male children) | 2-4 years
  Measured by orichodometer in milimeters.
Anogenital distance (AGD) (male and female children) | 2-4 years
  Distance from anus to genital tubercle, measured in milimeters with a caliper
Penile measurements (male children) | 2-4 years
  Penile measurements with a caliper measured in milimeters
Assessment Palpable Breast Tissue in female participants | 2-4 years
  Breast development will be assessed by palpation. The presence or absence of palpable breast tissue will be recorded. If present, the diameter will also be measured in millimeters using a ruler.
Assessment of Tanner stages (male and female children) | 2-4 years
  Assessment of pubic hair development, and staging it according to the tanner stages.
DNA methylation patterns (male and female children) | 2-4 years
  DNA methylation patterns will be analyzed with the Illumina Infinium MethylationEPIC v2.0 BeadChip.
Presence of Selected Genetic Variants Related to Hormone Regulation -Targeted SNP analyses (male and female children) | 2-4 years
  Targeted SNP analysis will be performed on a predefined set of genetic polymorphisms (up to 200 genes) associated with hormone production and receptor sensitivity. Analyses will be conducted using PCR genotyping or targeted sequencing. Whole-exome or genome-wide sequencing will not be performed, in accordance with Danish National Ethics Committee guidelines.
Urine sample (male and female children) | 2-4 years
  LH measured in IU/L using immunoassays
Urine sample (male and female children) | 2-4 years
  Endocrine disrupting chemical: phthalates using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Urine sample (male and female children) | 2-4 years
  Endocrine disrupting chemical: phenols using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Urine sample (male and female children) | 2-4 years
  Endocrine disrupting chemical:, perfluorinated compounds using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Urine sample (male and female children) | 2-4 years
  Endocrine disrupting chemical: parabens using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Urine sample (male and female children) | 2-4 years
  Steroid hormone metabolites will be assessed in nmol/L using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Plasma serotonin (male and female children) | 2-4 years
  Plasma serotonin measured in ng/ml by using tandem massespektrometri

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Holm JB, Mazaud-Guittot S, Danneskiold-Samsoe NB, Chalmey C, Jensen B, Norregard MM, Hansen CH, Styrishave B, Svingen T, Vinggaard AM, Koch HM, Bowles J, Koopman P, Jegou B, Kristiansen K, Kristensen DM. Intrauterine Exposure to Paracetamol and Aniline Impairs Female Reproductive Development by Reducing Follicle Reserves and Fertility. Toxicol Sci. 2016 Mar;150(1):178-89. doi: 10.1093/toxsci/kfv332. Epub 2016 Jan 5. PMID 26732887
- [Background] Dean A, van den Driesche S, Wang Y, McKinnell C, Macpherson S, Eddie SL, Kinnell H, Hurtado-Gonzalez P, Chambers TJ, Stevenson K, Wolfinger E, Hrabalkova L, Calarrao A, Bayne RA, Hagen CP, Mitchell RT, Anderson RA, Sharpe RM. Analgesic exposure in pregnant rats affects fetal germ cell development with inter-generational reproductive consequences. Sci Rep. 2016 Jan 27;6:19789. doi: 10.1038/srep19789. PMID 26813099
- [Background] Bauer AZ, Swan SH, Kriebel D, Liew Z, Taylor HS, Bornehag CG, Andrade AM, Olsen J, Jensen RH, Mitchell RT, Skakkebaek NE, Jegou B, Kristensen DM. Paracetamol use during pregnancy - a call for precautionary action. Nat Rev Endocrinol. 2021 Dec;17(12):757-766. doi: 10.1038/s41574-021-00553-7. Epub 2021 Sep 23. PMID 34556849
- [Background] Rebordosa C, Kogevinas M, Bech BH, Sorensen HT, Olsen J. Use of acetaminophen during pregnancy and risk of adverse pregnancy outcomes. Int J Epidemiol. 2009 Jun;38(3):706-14. doi: 10.1093/ije/dyp151. Epub 2009 Mar 30. PMID 19332503
- [Background] Lind DV, Main KM, Kyhl HB, Kristensen DM, Toppari J, Andersen HR, Andersen MS, Skakkebaek NE, Jensen TK. Maternal use of mild analgesics during pregnancy associated with reduced anogenital distance in sons: a cohort study of 1027 mother-child pairs. Hum Reprod. 2017 Jan;32(1):223-231. doi: 10.1093/humrep/dew285. Epub 2016 Nov 16. PMID 27852690
- [Background] Ersboll AS, Hedegaard M, Damm P, Johansen M, Tabor A, Hegaard HK. Changes in the pattern of paracetamol use in the periconception period in a Danish cohort. Acta Obstet Gynecol Scand. 2015 Aug;94(8):898-903. doi: 10.1111/aogs.12667. Epub 2015 May 29. PMID 25939806
- [Background] Kristensen DM, Mazaud-Guittot S, Gaudriault P, Lesne L, Serrano T, Main KM, Jegou B. Analgesic use - prevalence, biomonitoring and endocrine and reproductive effects. Nat Rev Endocrinol. 2016 Jul;12(7):381-93. doi: 10.1038/nrendo.2016.55. Epub 2016 May 6. PMID 27150289
- [Background] Roberge S, Bujold E, Nicolaides KH. Aspirin for the prevention of preterm and term preeclampsia: systematic review and metaanalysis. Am J Obstet Gynecol. 2018 Mar;218(3):287-293.e1. doi: 10.1016/j.ajog.2017.11.561. Epub 2017 Nov 11. PMID 29138036
- [Background] Cadavid AP. Aspirin: The Mechanism of Action Revisited in the Context of Pregnancy Complications. Front Immunol. 2017 Mar 15;8:261. doi: 10.3389/fimmu.2017.00261. eCollection 2017. PMID 28360907
- [Background] Nitsche JF, Patil AS, Langman LJ, Penn HJ, Derleth D, Watson WJ, Brost BC. Transplacental Passage of Acetaminophen in Term Pregnancy. Am J Perinatol. 2017 May;34(6):541-543. doi: 10.1055/s-0036-1593845. Epub 2016 Nov 2. PMID 27806383
- [Background] Koehn L, Habgood M, Huang Y, Dziegielewska K, Saunders N. Determinants of drug entry into the developing brain. F1000Res. 2019 Aug 7;8:1372. doi: 10.12688/f1000research.20078.1. eCollection 2019. PMID 31656590
- [Background] Olesen TS, Bleses D, Andersen HR, Grandjean P, Frederiksen H, Trecca F, Bilenberg N, Kyhl HB, Dalsager L, Jensen IK, Andersson AM, Jensen TK. Prenatal phthalate exposure and language development in toddlers from the Odense Child Cohort. Neurotoxicol Teratol. 2018 Jan-Feb;65:34-41. doi: 10.1016/j.ntt.2017.11.004. Epub 2017 Dec 1. PMID 29198963
- [Background] Hansen JB, Bilenberg N, Timmermann CAG, Jensen RC, Frederiksen H, Andersson AM, Kyhl HB, Jensen TK. Prenatal exposure to bisphenol A and autistic- and ADHD-related symptoms in children aged 2 and5 years from the Odense Child Cohort. Environ Health. 2021 Mar 12;20(1):24. doi: 10.1186/s12940-021-00709-y. PMID 33712018
- [Background] Guilbert A, Rolland M, Pin I, Thomsen C, Sakhi AK, Sabaredzovic A, Slama R, Guichardet K, Philippat C. Associations between a mixture of phenols and phthalates and child behaviour in a French mother-child cohort with repeated assessment of exposure. Environ Int. 2021 Nov;156:106697. doi: 10.1016/j.envint.2021.106697. Epub 2021 Jun 18. PMID 34147998
- [Background] Arendrup FS, Mazaud-Guittot S, Jegou B, Kristensen DM. EDC IMPACT: Is exposure during pregnancy to acetaminophen/paracetamol disrupting female reproductive development? Endocr Connect. 2018 Jan;7(1):149-158. doi: 10.1530/EC-17-0298. Epub 2018 Jan 5. PMID 29305399
- [Background] Kristensen DM, Hass U, Lesne L, Lottrup G, Jacobsen PR, Desdoits-Lethimonier C, Boberg J, Petersen JH, Toppari J, Jensen TK, Brunak S, Skakkebaek NE, Nellemann C, Main KM, Jegou B, Leffers H. Intrauterine exposure to mild analgesics is a risk factor for development of male reproductive disorders in human and rat. Hum Reprod. 2011 Jan;26(1):235-44. doi: 10.1093/humrep/deq323. Epub 2010 Nov 8. PMID 21059752
- [Background] Reel JR, Lawton AD, Lamb JC 4th. Reproductive toxicity evaluation of acetaminophen in Swiss CD-1 mice using a continuous breeding protocol. Fundam Appl Toxicol. 1992 Feb;18(2):233-9. doi: 10.1016/0272-0590(92)90051-i. PMID 1601223
- [Background] Johansson HK, Jacobsen PR, Hass U, Svingen T, Vinggaard AM, Isling LK, Axelstad M, Christiansen S, Boberg J. Perinatal exposure to mixtures of endocrine disrupting chemicals reduces female rat follicle reserves and accelerates reproductive aging. Reprod Toxicol. 2016 Jun;61:186-94. doi: 10.1016/j.reprotox.2016.03.045. Epub 2016 Apr 2. PMID 27049580
- [Background] Hurtado-Gonzalez P, Anderson RA, Macdonald J, van den Driesche S, Kilcoyne K, Jorgensen A, McKinnell C, Macpherson S, Sharpe RM, Mitchell RT. Effects of Exposure to Acetaminophen and Ibuprofen on Fetal Germ Cell Development in Both Sexes in Rodent and Human Using Multiple Experimental Systems. Environ Health Perspect. 2018 Apr 16;126(4):047006. doi: 10.1289/EHP2307. PMID 29665328
- [Background] Wolf C Jr, Lambright C, Mann P, Price M, Cooper RL, Ostby J, Gray LE Jr. Administration of potentially antiandrogenic pesticides (procymidone, linuron, iprodione, chlozolinate, p,p'-DDE, and ketoconazole) and toxic substances (dibutyl- and diethylhexyl phthalate, PCB 169, and ethane dimethane sulphonate) during sexual differentiation produces diverse profiles of reproductive malformations in the male rat. Toxicol Ind Health. 1999 Jan-Mar;15(1-2):94-118. doi: 10.1177/074823379901500109. PMID 10188194
- [Background] Drake AJ, van den Driesche S, Scott HM, Hutchison GR, Seckl JR, Sharpe RM. Glucocorticoids amplify dibutyl phthalate-induced disruption of testosterone production and male reproductive development. Endocrinology. 2009 Nov;150(11):5055-64. doi: 10.1210/en.2009-0700. Epub 2009 Oct 9. PMID 19819957
- [Background] Holm JB, Chalmey C, Modick H, Jensen LS, Dierkes G, Weiss T, Jensen BA, Norregard MM, Borkowski K, Styrishave B, Martin Koch H, Mazaud-Guittot S, Jegou B, Kristiansen K, Kristensen DM. Aniline Is Rapidly Converted Into Paracetamol Impairing Male Reproductive Development. Toxicol Sci. 2015 Nov;148(1):288-98. doi: 10.1093/toxsci/kfv179. Epub 2015 Aug 10. PMID 26259604
- [Background] Nielsen JK, Modick H, Morck TA, Jensen JF, Nielsen F, Koch HM, Knudsen LE. N-acetyl-4-aminophenol (paracetamol) in urine samples of 6-11-year-old Danish school children and their mothers. Int J Hyg Environ Health. 2015 Jan;218(1):28-33. doi: 10.1016/j.ijheh.2014.07.001. Epub 2014 Jul 24. PMID 25127489
- [Background] Bleses D, Vach W, Slott M, Wehberg S, Thomsen P, Madsen TO, Basboll H. The Danish Communicative Developmental Inventories: validity and main developmental trends. J Child Lang. 2008 Aug;35(3):651-69. doi: 10.1017/S0305000907008574. PMID 18588718
- [Background] Fenson L, Marchman VA, Thal DJ, Dale PS, Reznick JS, Bates E. MacArthur-Bates Communicative Development Inventories: User's Guide and Technical Manual (2nd ed.) 2007; Baltimore, MD: Brookes.
- [Background] Golombok S, Rust J. The Pre-School Activities Inventory: A standardized assessment of gender role in children. Psychol Assess. 1993 Jun;5(2):131-6.
- [Background] Kristensen S, Henriksen TB, Bilenberg N. The Child Behavior Checklist for Ages 1.5-5 (CBCL/1(1/2)-5): assessment and analysis of parent- and caregiver-reported problems in a population-based sample of Danish preschool children. Nord J Psychiatry. 2010 May 4;64(3):203-9. doi: 10.3109/08039480903456595. PMID 20085433
- [Background] Peric M, Beceheli I, Cicin-Sain L, Desoye G, Stefulj J. Serotonin system in the human placenta - the knowns and unknowns. Front Endocrinol (Lausanne). 2022 Dec 1;13:1061317. doi: 10.3389/fendo.2022.1061317. eCollection 2022. PMID 36531448
- [Background] Marotta R, Risoleo MC, Messina G, Parisi L, Carotenuto M, Vetri L, Roccella M. The Neurochemistry of Autism. Brain Sci. 2020 Mar 13;10(3):163. doi: 10.3390/brainsci10030163. PMID 32182969
- [Background] Barbosa AG, Pratesi R, Paz GSC, Dos Santos MAAL, Uenishi RH, Nakano EY, Gandolfi L, Pratesi CB. Assessment of BDNF serum levels as a diagnostic marker in children with autism spectrum disorder. Sci Rep. 2020 Oct 15;10(1):17348. doi: 10.1038/s41598-020-74239-x. PMID 33060610
- [Background] Polacchini A, Metelli G, Francavilla R, Baj G, Florean M, Mascaretti LG, Tongiorgi E. A method for reproducible measurements of serum BDNF: comparison of the performance of six commercial assays. Sci Rep. 2015 Dec 10;5:17989. doi: 10.1038/srep17989. PMID 26656852
- [Background] Rifas-Shiman SL, Cardenas A, Hivert MF, Tiemeier H, Bertoldi AD, Oken E. Associations of prenatal or infant exposure to acetaminophen or ibuprofen with mid-childhood executive function and behaviour. Paediatr Perinat Epidemiol. 2020 May;34(3):287-298. doi: 10.1111/ppe.12596. Epub 2019 Oct 21. PMID 31637744